CLINICAL TRIAL: NCT03172663
Title: Effect of Increased Body Mass Index on Auditory Function
Brief Title: Body Mass Index and Audiology Function
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, NElshreef, principal investigator, Assiut University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: AUDIO
Record Dates: First submitted 2017-05-26; First posted 2017-06-01 (Actual); Last update posted 2017-06-06 (Actual); Status verified 2017-05

CONDITIONS: Hearing Loss
Keywords: obesity
MeSH Terms: conditions — Hearing Loss; Obesity | interventions — Audiometry, Pure-Tone

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group 1 (Experimental)
  Interventions: Device: pure tone audiometry
- group 2 (Active Comparator)
  Interventions: Device: pure tone audiometry

INTERVENTIONS:
Device: pure tone audiometry — for estimate the type and degree of hearing loss

SUMMARY:
Obesity may directly or indirectly lead to hearing loss

DETAILED DESCRIPTION:
Obesity is measured by Body Mass Index.it is calculated by dividing a person's weight in kilograms by the square of height in meters. For children and adolescent. Overweight is defined as Body Mass Index is <85th percentile <95th percentile but obesity is defined as body mass index at or above the 95th percentile for children and teens of the same age and sex the increasing in body mass index mass may affect auditory function Directly as adipose tissue secretes hormones and cytokines, proinflammatory cytokines lead to release of obesity-induced inflammation which may directly contribute to end-organ damage Also, Adiponectin, which is thought to have anti-inflammatory and antiatherogenic effects, and associated with favorable lipoprotein profile, independent of BMI and insulin resistance, low plasma concentrations of adiponectin have been associated with obesity in children. In adults, low level of adiponectin has been associated with elevated high-frequency thresholds.

Indirectly, by obesity comorbidities including Hypertension, Type 2 diabetes mellitus, Dyslipidemia , Metabolic Syndrome and Cardiovascular Diseases

ELIGIBILITY:
Inclusion Criteria:

It will include 50 subjects whose:

* Age ranges from 10 to 40 years old.
* Body Mass Index more than the 85th percentile.
* male and female will be included

Exclusion Criteria:

* External or middle ear disease that causes conductive hearing loss such as otitis media, otomycosis, perforated drum, tumors, dislocation of the ossicles.
* High environmental noise exposure which causes acoustic trauma such as exploration, fire shots and noise in industries.
* ototoxic drug intake such as Aspirin, Aminoglycosides, Erythromycin, Vancomycin Streptomycin, Kanamycin, Neomycin, Gentamycin, Tobramycin, Lasix, Cisplatin, Nitrogen Mustard, and Vincristine, and Quinine.
* Major neurological or psychiatric diseases brain tumor, vestibular Schwannoma, stroke, acoustic neuroma, encephalitis, meningitis, and depression.

Ages: 10 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-05-01 (Estimated); Primary Completion 2019-05-01 (Estimated); Study Completion 2019-11-01 (Estimated)

PRIMARY OUTCOMES:
body mass index | 20 minutes
  if increased body mass index affect auditory function assessed by pure tone audiomertry

REFERENCES:
- [Background] Ogden CL, Carroll MD, Kit BK, Flegal KM. Prevalence of obesity and trends in body mass index among US children and adolescents, 1999-2010. JAMA. 2012 Feb 1;307(5):483-90. doi: 10.1001/jama.2012.40. Epub 2012 Jan 17. PMID 22253364